CLINICAL TRIAL: NCT01227356
Title: A Randomized Study Comparing Imatinib And Imatinib/Pegylated Interferon Alpha-2B in Newly Diagnosed Non-high Risk Chronic Myeloid Leukemia Patients in Complete Hematological Remission After Imatinib Induction Therapy
Brief Title: A Study Comparing Imatinib and Imatinib/Pegylated Interferon in Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Bengt Simonsson/Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NordCML002
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Health Care Quality; Health Care Evaluation
Keywords: Chronic myeloid leukemia, imatinib, interferon
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imatinb + pegIntron (Experimental)
  Interventions: Drug: imatinib and pegylated interferon

INTERVENTIONS:
Drug: imatinib and pegylated interferon — imatinib 400 mg p.o. daily pegylated interferon 50 ug s.c. weekly
  Other Names: Gleevec; PegIntron

SUMMARY:
Patients with chronic myeloid leukemia in imatinib induced CHR are randomized between imatinib 400 mg daily and imatinib 400 mg daily + PegIntron 30 ug weekly.

Primary endpoint: To compare at 12 months between the treatment arms the rate of Major Molecular Response (=99,9% tumour reduction) at 12 months

DETAILED DESCRIPTION:
130 patients registered, 112 randomized. 56 pats in each treatment arm. 12 months study duration. Rate of Major Molecular Response was at 12 months 53 vs 82 % (p=0.002) in favour of the combination arm.

ELIGIBILITY:
Inclusion Criteria:

Chronic myeloid leukemia in imatinib induced complete hematological remission. Intermediate/low risk, ECOG < 2

Exclusion Criteria:

Les than CHR after 3 months imatinib high risk More than 6 months from diagnosis ECOG > 2 Pregnancy

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-09; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Comparison of rate Major Molecular Response between treatment arms | 2004 - 2009
  Molecular response

SECONDARY OUTCOMES:
Comparison of complete cytogenetic response between the treatment arms at 12 months | 2004 - 2009
  Cytogenetic response
Comparison rate complete cytogenetic response between the treatment arms at 12 months | 2004 - 2009
  Hematologic response

CONTACTS AND LOCATIONS:
Overall Officials: bengt NO Simonsson, MD, PhD, Study Chair — Uppsala University
Locations (2):
- Sweden (2):
  - Bengt Simonsson, Uppsala
  - Uppsala University Hospital, Uppsala